CLINICAL TRIAL: NCT04058353
Title: A Phase 3, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445 Combination Therapy in Subjects With Cystic Fibrosis Who Are Heterozygous for the F508del Mutation and a Gating or Residual Function Mutation (F/G and F/RF Genotypes)
Brief Title: A Phase 3 Study of VX-445 Combination Therapy in Cystic Fibrosis (CF) Subjects Heterozygous for F508del and a Gating or Residual Function Mutation (F/G and F/RF Genotypes)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX18-445-104; 2018-002835-76 (EudraCT Number)
Expanded Access: NCT04058210 (Approved for marketing)
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor; tezacaftor, ivacaftor drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control: IVA or TEZ/IVA (Active Comparator): Following an IVA or TEZ/IVA run-in period of 4 weeks, participants either received IVA 150 milligrams (mg) every 12 hours (q12h) or TEZ 100 mg once daily (qd)/IVA 150 mg q12h in the treatment period for 8 weeks.
  Interventions: Drug: IVA; Drug: TEZ/IVA
- TC: ELX/TEZ/IVA (Experimental): Following an IVA or TEZ/IVA run-in period of 4 weeks, participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 8 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — FDC tablet for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
  Arms: TC: ELX/TEZ/IVA
Drug: IVA — Mono-tablet for oral administration.
  Other Names: VX-770; ivacaftor
Drug: TEZ/IVA — Fixed-dose combination (FDC) tablet for oral administration.
  Other Names: VX-661/VX-770; tezacaftor/ivacaftor
  Arms: Control: IVA or TEZ/IVA

SUMMARY:
This study will evaluate the efficacy, safety and pharmacodynamics of elexacaftor (ELX, VX-445) in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are heterozygous for F508del and a gating or residual function mutation (F/G and F/RF genotypes).

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has a confirmed diagnosis of CF and is heterozygous for F508del and either a gating or residual function mutation (F/G and F/RF genotypes)
* Forced expiratory volume in 1 second (FEV1) value ≥40% and ≤90% of predicted mean for age, sex, and height

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (93):
- United States (37):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Miller Children's Hospital / Long Beach Memorial, Long Beach, California
  - Stanford University, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco, Lung Transplant Program, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Indiana University, Indianapolis, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital Cystic Fibrosis Center Clinical Rsearch Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Northwell Health- Long Island Jewish Medical Center, New Hyde Park, New York
  - Mount Sinai Beth Israel, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - UC Health Holmes, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - ProMedica Toledo Hospital/Toledo Children's Hospital/Pediatric Pulmonary & Cystic Fibrosis Center, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Dell Children's Medical Group, Austin, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah / Primary Children's Medical Center, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (7):
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne, VIC
  - Perth Children's Hospital, Nedlands
  - The Royal Children's Hospital, Parkville, VIC
  - Mater Adult Hospital, South Brisbane
  - Queensland Children's Hospital, South Brisbane
  - Westmead Hospital, Westmead
- Belgium (4):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (4):
  - Stollery Children's Hospital, Edmonton
  - McGill University Health Center, Québec
  - St. Michael's Hospital, Toronto
  - St. Paul's Hospital, Vancouver
- Juliane Marie Center, Rigshospitalet, Copenhagen, Denmark
- France (8):
  - Centre Hospitalier Lyon Sud, Benite Cedex
  - Groupe Hospitaler Pellegrin, CHU De Bordeaux, Bordeaux
  - CHRU de Lille - Hopital Albert Calmette, Lille
  - CHU Marseille - Hopital Nord, Marseille
  - CHU de Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - Hopital Cochin, Paris
  - Hopital Necker, Enfants Malades, Paris
  - Hopital Pontchaillou CHU de Rennes, Rennes
- Germany (7):
  - Charite Paediatric Pulmonology Department, Berlin
  - Friedrich-Alexander University of Erlangen-Nuremberg, University Children's Hospital, Erlangen
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Justus-Liebig-Universitaet Gießen Zentrum fur Kinderheilkunde und Jugendmedizin, Giessen
  - Universitätsklinikum Halle (Saale) / Universitätsklinik und Poliklinik für Innere Medizin, Schwerpunkt Pneumologie, Halle
  - Pneumologisches Studienzentrum Muenchen-West, München
  - University Hospital Wuerzburg, Würzburg
- Ireland (3):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
- University Hospital Limerick (Adults), Limerick, Israel
- Italy (6):
  - Azienda Ospedaliero Universitaria Ospedale Riuniti, Ancona
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Malattie Apparato Respiratorio 2 - Fibrosi Cistica, Orbassano
  - Ospedale Pediatrico Bambino Gesu, Rome
  - Azienda Ospedaliera di Verona-Ospedale Civile Maggiore, Verona
- Netherlands (3):
  - University Medical Center, Utrecht, Department of Pulmonology and Tuberculosis, Heidelberglaan
  - UMC St. Radboud, Nijmegen
  - HagaZiekenhuis van den Haag, The Hague
- Spain (4):
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- United Kingdom (8):
  - Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge
  - Royal Devon and Exeter NHS Foundation Trust, Royal Devon and Exeter Hospital, Exeter
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - St. James University Hospital, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Wythenshawe Hospital, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Barry PJ, Mall MA, Alvarez A, Colombo C, de Winter-de Groot KM, Fajac I, McBennett KA, McKone EF, Ramsey BW, Sutharsan S, Taylor-Cousar JL, Tullis E, Ahluwalia N, Jun LS, Moskowitz SM, Prieto-Centurion V, Tian S, Waltz D, Xuan F, Zhang Y, Rowe SM, Polineni D; VX18-445-104 Study Group. Triple Therapy for Cystic Fibrosis Phe508del-Gating and -Residual Function Genotypes. N Engl J Med. 2021 Aug 26;385(9):815-825. doi: 10.1056/NEJMoa2100665. PMID 34437784

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 271 participants were enrolled in this study out of which 12 participants discontinued in run-in period. Of 259 participants, 1 participant was randomized but not dosed in the treatment period. Therefore, results are presented for only 258 participants.
Pre-assignment Details: This study was conducted in cystic fibrosis (CF) participants aged 12 years or older.
Groups:
- Control: IVA or TEZ/IVA: Following an IVA (ivacaftor) or TEZ (tezacaftor)/IVA run-in period of 4 weeks, participants either received IVA 150 milligrams (mg) every 12 hours (q12h) or TEZ 100 mg once daily (qd)/IVA 150 mg q12h in the treatment period for 8 weeks.
- Triple Combination (TC): ELX/TEZ/IVA: Following an IVA or TEZ/IVA run-in period of 4 weeks, participants received ELX (elexacaftor) 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 8 weeks.
Period: Overall Study
Arm/Group | Control: IVA or TEZ/IVA | Triple Combination (TC): ELX/TEZ/IVA
Started | 126 | 132
Completed | 122 | 131
Not Completed | 4 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: IVA or TEZ/IVA: Following an IVA or TEZ/IVA run-in period of 4 weeks, participants either received IVA 150 mg q12h or TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Control: IVA or TEZ/IVA | TC: ELX/TEZ/IVA | Total
Number analyzed (Participants) | 126 | 132 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (14.3) | 37.7 (14.7) | 37.7 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 67 | 128
  Male | 65 | 65 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 114 | 117 | 231
  Unknown or Not Reported | 8 | 10 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 0 | 2
  Not Collected per Local Regulations | 9 | 9 | 18
  Aboriginal | 2 | 1 | 3
  Latin-American | 1 | 0 | 1
  Lebanese | 1 | 0 | 1
  White | 110 | 122 | 232
  White, American Indian or Alaska Native | 1 | 0 | 1
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) [Mean (Standard Deviation); unit: percentage points] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  percentage points | 68.1 (16.4) | 67.1 (15.7) | 67.6 (16.0)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) for ELX/TEZ/IVA Group
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Week 8
Population: Full analysis set (FAS) included all randomized participants who have the intended CF transmembrane conductance regulator (CFTR) allele mutation and received at least 1 dose of study drug in the treatment period. This outcome measure was applicable only for the triple combination arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | TC: ELX/TEZ/IVA
Number analyzed (Participants) | 132
percentage points | 3.7 [2.8 to 4.6]

2. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl) for ELX/TEZ/IVA Group
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 8
Population: FAS. This outcome measure was applicable only for the triple combination group.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per Liter (mmol/L)
Arm/Group | TC: ELX/TEZ/IVA
Number analyzed (Participants) | 132
millimole per Liter (mmol/L) | -22.3 [-24.5 to -20.2]

3. Secondary Outcome: Absolute Change in ppFEV1 for the ELX/TEZ/IVA Group Compared to the Control Group
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Week 8
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage points
Arm/Group | Control: IVA or TEZ/IVA | TC: ELX/TEZ/IVA
Number analyzed (Participants) | 126 | 132
percentage points | 0.2 [-0.7 to 1.1] | 3.7 [2.8 to 4.6]
Statistical Analysis 1: Comparison: Control: IVA or TEZ/IVA vs TC: ELX/TEZ/IVA; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; Least Squares (LS) Mean Difference = 3.5, 95% CI 2-sided [2.2 to 4.7]

4. Secondary Outcome: Absolute Change in SwCl for ELX/TEZ/IVA Group Compared to the Control Group
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 8
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Control: IVA or TEZ/IVA | TC: ELX/TEZ/IVA
Number analyzed (Participants) | 126 | 132
mmol/L | 0.7 [-1.4 to 2.8] | -22.3 [-24.5 to -20.2]
Statistical Analysis 1: Comparison: Control: IVA or TEZ/IVA vs TC: ELX/TEZ/IVA; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = -23.1, 95% CI 2-sided [-26.1 to -20.1]

5. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score for ELX/TEZ/IVA Group
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline Through Week 8
Population: FAS. This outcome measure was applicable only for the triple combination arm.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TC: ELX/TEZ/IVA
Number analyzed (Participants) | 132
units on a scale | 10.3 [8.0 to 12.7]

6. Secondary Outcome: Absolute Change in CFQ-R Respiratory Domain Score for ELX/TEZ/IVA Group Compared to the Control Group
Description: as for outcome 5
Time Frame: From Baseline Through Week 8
Population: FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control: IVA or TEZ/IVA | TC: ELX/TEZ/IVA
Number analyzed (Participants) | 126 | 132
units on a scale | 1.6 [-0.8 to 4.1] | 10.3 [8.0 to 12.7]
Statistical Analysis 1: Comparison: Control: IVA or TEZ/IVA vs TC: ELX/TEZ/IVA; Test type: Superiority; p < 0.0001, Mixed-effects model for repeated measure; LS Mean Difference = 8.7, 95% CI 2-sided [5.3 to 12.1]

7. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 12
Population: Safety set included all participants who received at least 1 dose of study drug in the treatment period.
Measure: Number; unit: participants
Arm/Group | Control: IVA or TEZ/IVA | TC: ELX/TEZ/IVA
Number analyzed (Participants) | 126 | 132
participants
  Participants With TEAEs | 83 | 88
  Participants With SAEs | 11 | 5

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 12
Arm/Group | Control: IVA or TEZ/IVA | TC: ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/132
Serious Adverse Events (participants affected / at risk) | 11/126 | 5/132
Other Adverse Events (participants affected / at risk) | 47/126 | 35/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control: IVA or TEZ/IVA (N=126) | TC: ELX/TEZ/IVA (N=132)
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 7 | 2
Pneumonia (Infections and infestations) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control: IVA or TEZ/IVA (N=126) | TC: ELX/TEZ/IVA (N=132)
Abdominal pain (Gastrointestinal disorders) | 2 | 7
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Nausea (Gastrointestinal disorders) | 9 | 2
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 10 | 2
Alanine aminotransferase increased (Investigations) | 0 | 8
Aspartate aminotransferase increased (Investigations) | 0 | 8
Headache (Nervous system disorders) | 19 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 3
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT04058353/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT04058353/SAP_001.pdf